CLINICAL TRIAL: NCT04467359
Title: Application of Rapid Rehabilitation Nursing in Perioperative Rehabilitation of Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018180520
Record Dates: First submitted 2020-06-28; First posted 2020-07-13 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2020-10

CONDITIONS: Knee Arthroscopy
Keywords: Nursing; Enhanced Recovery After Surgery（ERAS）

STUDY DESIGN:
Intervention Model Description: The subjects were randomly divided into the experimental group and the control group. The control group received conventional rehabilitation nursing during the perioperative period, while the experimental group received ERAS intervention. The differences between the two groups in postoperative pain degree (NRS0-10) comfort level (Likert 1-5) and rehabilitation completion Range of motion(ROM) score were compared. The safety index was the occurrence of postoperative complications such as nausea, vomiting, dizziness, headache and urinary retention, and the occurrence of postoperative complications such as hypothermia after lower extremity deep venous thrombosis (preoperative and postoperative comparison of ESR CRP and procalcitonin indexes in blood routine)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group (Experimental): ERAS intervention group
  Interventions: Other: ERAS; Other: Perioperative routine rehabilitation nursing
- The control group (Placebo Comparator): Sports medicine rehabilitation nursing group
  Interventions: Other: Perioperative routine rehabilitation nursing

INTERVENTIONS:
Other: ERAS — Optimize physical conditions; Fasting solid diet 6h before surgery, fasting clear fluid 2 h before surgery; If there is no chief complaint of dizziness, nausea or other discomfort after the operation, warm water (no more than 100ml) can be immediately drunk. Pain management; Encourage patients to engage in early activities under the premise of effective pain control; If no dural puncture and other complications occur, the patient has no chief complaints of headache, dizziness, nausea and other discomfort, and there is no need to lie supine, the comfortable position such as semi-supine lateral supine position can be taken immediately (avoid 90-degree upright position for patients with hip joint); Prevention of thrombosis; Prevention and treatment of nausea and vomiting; Follow-up was conducted at 4 weeks, 8 weeks and 12 weeks after the operation.
  Arms: The experimental group
Other: Perioperative routine rehabilitation nursing — Fasting and water deprivation at 12 o 'clock on the first day before surgery; Fasting water 6-8 hours after surgery; Lie flat on your pillow for 6 hours; Get out of bed activity 1 day after operation

SUMMARY:
The purpose of this study is to apply the concept of rapid rehabilitation nursing in the perioperative period of knee arthroscopy, to make up for the gap in this field, to provide reference basis for the general colleagues, promote the development of perioperative rapid rehabilitation nursing of knee arthroscopy, accelerate the rehabilitation of patients.

DETAILED DESCRIPTION:
This study aims to apply rapid rehabilitation nursing concept to the arthroscopic perioperative nursing, used to make up for the blank in this field, provides the reference for the overwhelming majority of peer, prompt the arthroscopic perioperative rehabilitation nursing development, accelerate the patient rehabilitation in January 2020 - December 2020 in Beijing a third rate sports medicine hospital be in hospital, to line the arthroscopic surgery patients as the research object, adopt the method of prospective, randomized, controlled in 220 patients. Inclusion criteria: < 60 age 18 years old, patients with informed consent and voluntary participation in arthroscopic anterior cruciate ligament reconstruction under external anesthesia were excluded from this study: patients with mental system diseases or communication disorders; Patients with metabolic diseases such as diabetes; Patients who could not quit smoking and drinking alcohol before surgery as required; Patients with gastrointestinal tract disease research object were randomly divided into experimental group and control group, control group given conventional perioperative nursing, the experimental group to implement rapid rehabilitation program, the specific implementation process, see table 1 and table 2, compare two groups of preoperative postoperative self-care ability score (Barthel index) 、 the degree of postoperative pain numerical rating scale (NRS 0-10 score) 、the degree of comfort (Likert 1-5 rating score) and rehabilitation completion -Range of motion(ROM) score difference; The safety index was the occurrence of postoperative complications such as nausea, vomiting, dizziness, headache and urinary retention, and the occurrence of postoperative complications such as hypothermia after lower extremity deep venous thrombosis (preoperative and postoperative comparison of erythrocyte sedimentation rate(ESR)、C-reactive protein（CRP） and procalcitonin indexes in blood routine

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic anterior cruciate ligament reconstruction was performed under epidural anesthesia
* The patients consented and volunteered to participate in this study

Exclusion Criteria:

* Patients with mental disorders or communication disorders
* Patients with metabolic diseases such as diabetes
* Patients who could not quit smoking and drinking alcohol before surgery as required
* Patients with gastrointestinal disorders
* Patients who are not under epidural anesthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Self-care ability score | 1 day before operation
  Barthel Index:Barthel index is scored from 0 to 100. A score of 100 indicates that the patient has a good function in basic daily activities. He/she does not need help from others. He/she is able to control urine and urine, eat, dress, transfer to bed and chair, bathe, walk for at least one block, and can go up and down stairs. A score of 0 indicates poor functioning, lack of independence, and need help with all aspects of daily life. According to the score of Barthel index, the ability of daily activities was divided into three levels: good, medium and poor >. 60 was classified as good. 60 to 41 is medium. Have moderate dysfunction and need great help to complete daily activities; ≤40 is classified as poor, with severe dysfunction, most daily activities cannot be completed or need to be attended to by others.
Self-care ability score | Postoperative 1 day
  Barthel Index:Barthel index is scored from 0 to 100. A score of 100 indicates that the patient has a good function in basic daily activities. He/she does not need help from others. He/she is able to control urine and urine, eat, dress, transfer to bed and chair, bathe, walk for at least one block, and can go up and down stairs. A score of 0 indicates poor functioning, lack of independence, and need help with all aspects of daily life. According to the score of Barthel index, the ability of daily activities was divided into three levels: good, medium and poor >. 60 was classified as good. 60 to 41 is medium. Have moderate dysfunction and need great help to complete daily activities; ≤40 is classified as poor, with severe dysfunction, most daily activities cannot be completed or need to be attended to by others.
Degree of postoperative pain | Postoperative 1 day
  Numerical Rating Scale(NRS )score:0 means no pain, 10 means the most severe pain imaginable, and the higher the score, the more severe the pain
Comfort level | Postoperative 1 day
  Likert 1-5 score:0 means very uncomfortable, 10 means very comfortable, and the higher the score, the higher the comfort
Rehabilitation Completion | 2 weeks after discharged
  Range of motion(ROM):Use a square to measure the Angle of motion
Rehabilitation Completion | 4 weeks after discharged
  Range of motion(ROM):Use a square to measure the Angle of motion
Rehabilitation Completion | 8 weeks after discharged
  Range of motion(ROM):Use a square to measure the Angle of motion
Rehabilitation Completion | 12 weeks after discharged
  Range of motion(ROM):Use a square to measure the Angle of motion

SECONDARY OUTCOMES:
adverse reaction | postoperative 1 day
  Postoperative nausea, vomiting, dizziness, headache, urinary retention and other non-reaction occurred

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking Universitu 3rd Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No